CLINICAL TRIAL: NCT01798953
Title: Ileal Pouch-anal Anastomosis or Ileo-rectal Anastomosis for Patients With Ulcerative Colitis and Primary Sclerosing Cholangitis?
Brief Title: Surgical Reconstruction in Ulcerative Colitis With Primary Sclerosing Cholangitis
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Mattias Block, Doctor, Surgeon, MD, Sahlgrenska University Hospital
Other Study IDs: 326-10
Record Dates: First submitted 2013-02-19; First posted 2013-02-26 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Ulcerative Colitis; Primary Sclerosing Cholangitis; Pouchitis; Complications
Keywords: Ulcerative Colitis; Primary Sclerosing Cholangitis; Ileal pouch-anal anastomosis; Ileorectal anastomosis; Surgical outcome; Functional outcome; Failure
MeSH Terms: conditions — Colitis, Ulcerative; Cholangitis, Sclerosing; Pouchitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- UC/PSC with IPAA: Patients with ulcerative colitis and primary sclerosing cholangitis reconstructed with ileal pouch-anal anastomosis
- UC with IPAA: Patients with ulcerative colitis reconstructed with ileal pouch-anal anastomosis.
- UC/PSC with IRA: Patients with ulcerative colitis and primary sclerosing cholangitis reconstructed with ileorectal anastomosis.
- UC with IRA: Patients with ulcerative colitis reconstructed with ileorectal anastomosis.

SUMMARY:
Primary sclerosing cholangitis (PSC) occurs in approximately 10 % of patients with ulcerative colitis (UC), but the outcome of reconstructive surgery is not clear. The purpose of this study was to determine the functional outcome after surgery, frequency of pouchitis, complications and failure-rate in UC-PSC patients compared to patients with UC alone. Both ileal pouch-anal anastomosis (IPAA) and ileo-rectal anastomosis (IRA) were studied.

DETAILED DESCRIPTION:
Primary sclerosing cholangitis (PSC) is characterised by inflammation and fibrosis of the biliary tree and the condition can lead to end-stage liver disease. PSC is strongly associated with inflammatory bowel disease (IBD), with a prevalence of IBD in PSC as high as 60-84 % in Northern Europe and North America. The majority of patients with IBD and PSC have ulcerative colitis (UC).

Considering all patients with UC, around 30% will ultimately require surgery; the most common indications are acute colitis, chronic refractory disease or colorectal dysplasia. The standard procedure is proctocolectomy and ileal pouch-anal anastomosis (IPAA). However, ileo-rectal anastomosis (IRA) or conventional ileostomy are options. The prognosis after surgery is generally considered good.

Previous studies have shown that the course of colitis in patients with UC/PSC is different from that of patients with UC-only.

In a patient with UC, several aspects have to be considered at counselling before surgery. However, in many aspects, the literature is substantial for patients with UC-only (for example function and quality of life after IPAA) and key information can be safely provided. Conversely, patients with UC/PSC that require colectomy are rare and as a consequence, data on most aspects is sparse (18-20).

The aim of the study was to assess outcome after surgery (IPAA or IRA) in patients with UC/PSC. Focus was on pouch/rectal function, pouchitis, surgical complications and failure. Patients with UC-only were employed as controls.

ELIGIBILITY:
Inclusion Criteria:

* UC
* PSC
* IPAA
* IRA

Exclusion Criteria:

* non-UC
* non-PSC
* no consent

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with UC/PSC vs patients with UC only reconstructed surgically with IPAA or IRA.
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2010-01; Primary Completion 2013-02 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Functional outcome after reconstructive surgery with IPAA/IRA in patients with UC/PSC vs patients with UC only. | Up to six months

SECONDARY OUTCOMES:
Complications after reconstructive surgery with IPAA/IRA in patients with UC/PSC vs patients with UC only. | Up to six months.

OTHER OUTCOMES:
Failure after reconstructive surgery with IPAA/IRA in patients with UC/PSC vs patients with UC only. | Up to six months.

CONTACTS AND LOCATIONS:
Overall Officials: Lars G Börjesson, Ass Prof, Principal Investigator — Department of Surgery, Sahlgrenska, Göteborg
Locations (1):
- Department of Surgery, Inst for Clinical Sciences, Sahlgrenska University Hospital, Gothenburg, Göteborg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
PubMed